CLINICAL TRIAL: NCT07348627
Title: Opioid-Sparing Joint Replacement - Single Site Randomized Control Trial
Brief Title: Opioid-Sparing Joint Replacement
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ajay Premkumar, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025P011932
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Opioid Consumption
Keywords: Total hip arthroplasty; Numeric Rating Scale for pain; Visual Analog Scale for nausea; Life Care specialist
MeSH Terms: conditions — Agnosia | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-Sparing Regimen (Experimental): Participants receive a standardized multimodal non-opioid analgesic regimen throughout the perioperative period and are discharged with placebo tablets instead of a standard opioid prescription. All participants receive counseling from a Life Care Specialist and a limited supply of rescue hydromorphone for severe breakthrough pain.
  Interventions: Drug: Placebo; Other: Multimodal Non-Opioid Analgesia
- Standard Opioid Prescription (Active Comparator): Participants receive the same standardized multimodal non-opioid analgesic regimen and Life Care Specialist counseling as the experimental group, but are discharged with a standard opioid prescription.
  Interventions: Drug: Oxycodone 5 mg; Other: Multimodal Non-Opioid Analgesia

INTERVENTIONS:
Drug: Placebo — * 28 tablets identical in appearance to 5-mg oxycodone
  * Taken 1-2 tablets every 4 hours as needed for moderate to severe pain
  * Dispensed by Investigational Drug Services
  * Used in combination with standardized multimodal analgesia
  Arms: Opioid-Sparing Regimen
Drug: Oxycodone 5 mg — * 28 tablets of 5-mg oxycodone
  * Taken 1-2 tablets every 4 hours as needed for moderate to severe pain
  * Represents standard postoperative prescribing practi
  Arms: Standard Opioid Prescription
Other: Multimodal Non-Opioid Analgesia — Multimodal Non-Opioid Analgesia (Standardized Regimen)
  Includes:
  * Acetaminophen
  * Meloxicam
  * Methylprednisolone taper
  * Spinal anesthesia
  * Periarticular local anesthetic injection
  * Postoperative scheduled acetaminophen and NSAIDs
  * Counseling by Life Care Specialist
  * Two 2-mg hydromorphone tablets for rescue only

SUMMARY:
The goal of this clinical trial is to evaluate whether an opioid-sparing postoperative pain regimen can reduce opioid consumption and maintain effective pain control in adults undergoing anterior total hip arthroplasty for osteoarthritis.

The main questions it aims to answer are:

* Does an opioid-limited regimen result in lower postoperative opioid use compared with a standard opioid prescription?
* Does the opioid-limited regimen provide comparable or improved postoperative pain control and patient satisfaction?

DETAILED DESCRIPTION:
This study evaluates whether an opioid-sparing postoperative regimen can reduce opioid use while maintaining effective pain control in adults undergoing anterior total hip arthroplasty for osteoarthritis. Although opioids are commonly used after joint replacement, they carry risks such as side effects and long-term dependence. Multimodal analgesic strategies-using combinations of non-opioid medications and local anesthetic techniques-have shown promise in reducing opioid requirements while providing adequate pain relief.

All participants in this randomized, double-blind trial will receive a standardized multimodal non-opioid pain regimen throughout the perioperative period, along with counseling from a Life Care Specialist. Participants will be assigned to receive either a standard opioid prescription or placebo tablets at discharge, with a small supply of rescue hydromorphone available for severe breakthrough pain. Pain scores, nausea, opioid consumption, and patient-reported outcomes will be collected during the first postoperative week and at follow-up visits at 3 weeks and 3 months. The study aims to determine whether limiting routine opioid prescribing after hip arthroplasty can safely reduce opioid exposure without compromising recovery or patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hip osteoarthritis requiring primary arthroplasty
* Scheduled to undergo anterior total hip arthroplasty (THA)
* Able to comply with study procedures and follow-up visits
* Able to provide informed consent

Exclusion Criteria:

* Concurrent significant injuries to other bones or organs
* Local infection at or near the surgical site
* Preoperative opioid use within 4 weeks prior to surgery
* History of severe heart disease (NYHA Class II or higher), renal failure, or liver dysfunction
* Chronic liver disease
* Neurological or psychiatric conditions that may influence pain perception
* Pregnancy
* History of alcohol or medication abuse
* Inability to take NSAIDs
* Use of postoperative DVT prophylaxis other than aspirin 81 mg twice daily
* Diabetes mellitus with HbA1c > 8.0%
* Diagnosis of chronic pain syndrome or fibromyalgia
* Pain Catastrophizing Scale (PCS) score > 29
* Any condition that, in the investigator's judgment, may interfere with adherence to study procedures or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Daily Pain Scores (Numeric Rating Scale, NRS) | Postoperative Days 1-7
  A 0-10 numeric scale used to assess pain intensity. Participants rate their pain three times daily during the first postoperative week.
  Mean daily pain scores will be compared between groups. High scores: greater pain intensity. Low scores: better pain control.
Opioid Consumption (Morphine Milligram Equivalents, MME) | 1 week, 3 weeks, and 3 months postoperatively
  Total opioid use, including study medication, rescue hydromorphone, and any additional prescriptions, will be converted to MME to quantify postoperative opioid consumption.
Pain-Related Contacts to Clinical Team | Up to 3 months postoperatively
  Number of calls or electronic messages to the surgical team related to pain management.
Medication-Related Side Effects | Postoperative Days 1-7
  Incidence and severity of nausea, constipation, vomiting, or other adverse effects associated with postoperative pain medications.
Opioid Prescription Refills | Up to 3 months postoperatively
  Number of opioid prescription refills requested or obtained after surgery.
Patient Satisfaction With Pain Control | 1 week, 3 weeks, and 3 months
  Patient-reported satisfaction with postoperative pain control, rated on a 5-point scale (much worse than expected to much better than expected).

SECONDARY OUTCOMES:
Patient-Reported Outcomes (PROMs): HOOS Jr | Baseline (preoperative) and at 3 months
  Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS Jr.): A validated 6-item questionnaire assessing hip pain and functional ability in patients undergoing hip arthroplasty.
  0-100 (converted score)
  Interpretation:
  * Higher scores indicate better hip function and less pain.
  * Lower scores indicate greater disability or worse symptoms.
Patient-Reported Outcomes (PROMs): EQ-5D (EuroQol-5 Dimensions) | Baseline (preoperative) and at 3 months
  A standardized measure of health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Includes a health VAS.
  Index values typically 0-1 High scores: better overall health status. Low scores: poorer health or greater impairment.
Patient-Reported Outcomes (PROMs): Subjective Hip Value (SHV) | Baseline (preoperative) and at 3 months
  A single-item measure in which patients rate their hip function as a percentage of normal.
  * 0% = Completely nonfunctional hip
  * 100% = Completely normal hip
  Interpretation:
  * Higher percentages indicate better perceived hip function.
  * Lower percentages indicate worse perceived function.
Patient-Reported Outcomes (PROMs): Pain Catastrophizing Scale (PCS) | Baseline (preoperative) and at 3 months
  A 13-item questionnaire assessing catastrophic thinking related to pain (rumination, magnification, helplessness). Used at baseline for eligibility.
  Score range 0-52 High scores: greater pain catastrophizing; scores >29 indicate high catastrophizing. Low scores: minimal catastrophic thinking.
Postoperative Nausea (VAS-Nausea) | Postoperative Days 1-7
  Nausea severity recorded three times daily using a 0-10 Visual Analog Scale. A 0-10 scale used to measure severity of postoperative nausea. Recorded three times daily for 7 days.
  High scores: more severe nausea. Low scores: minimal or no nausea.
Sleep Quality and Pain-Related Satisfaction | Postoperative Days 1-7
  A patient-reported measure assessing perceived sleep quality and satisfaction with pain management during the study period.
  Both items use a 0-10 Numeric Rating Scale (NRS).
  * Higher scores indicate better sleep quality and greater satisfaction with pain management.
  * Lower scores indicate poorer sleep quality and lower satisfaction.
Length of Stay (LOS) | Day of surgery through discharge (usually upto 7 days)
  Duration of postoperative hospitalization.
Healthcare Utilization | Up to 3 months postoperatively
  Number of emergency department visits, readmissions, and reoperations related to the index surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Premkumar, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Orthopedics and Spine Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcomes of the study, including:
  Daily postoperative pain scores (Numeric Rating Scale, POD 1-7) Opioid consumption data (oral morphine equivalents) at 7 days, 3 weeks, and 3 months Patient-reported outcome measures (HOOS Jr., EQ-5D, Subjective Hip Value) Patient-reported satisfaction with pain control Medication-related side effects (e.g., nausea, constipation) Opioid refill information Length of stay, emergency department visits, readmissions, and reoperations
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after publication of the primary study results and will remain available for up to 5 years following publication, contingent upon institutional data retention policies.
Access Criteria: De-identified data will be shared with qualified researchers whose proposed use of the data has been approved by the study investigators.
  Requests for data access must be submitted to the corresponding author. Approved requests will be granted through a secure data-sharing mechanism (e.g., encrypted file transfer or institutional data-sharing platform) following execution of a data use agreement, as required.